CLINICAL TRIAL: NCT04971590
Title: LUNELORD: A Descriptive, Prospective Study to Assess Demographic, Pharmacologic, Biomarker, Clinical Features and QoL of Patients With LUpus NEphritis and Long-term ORgan Damage
Brief Title: Study to Assess Demographic, Pharmacologic, Biomarker, Clinical Features and Quality of Life (QoL) of Participants With Lupus Nephritis
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 216989
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: LUNELORD; Systemic lupus erythematosus; Lupus nephritis; Organ damage; Gulf countries; Real-world
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Lupus Nephritis
  Interventions: Other: Participant completed survey; Other: Medical chart review

INTERVENTIONS:
Other: Participant completed survey — Participants will be required to complete the participant survey.
Other: Medical chart review — Data will be collected from medical charts of participants.

SUMMARY:
This is a multicenter prospective study to assess clinical characteristics, demographics, treatment and health-related quality of life (HRQoL) of lupus nephritis (LN) participants across 5 Gulf countries (United Arab Emirates [UAE], Qatar, Bahrain, Kuwait and Oman).

ELIGIBILITY:
Inclusion Criteria:

* More than or equal to 18 years of age
* Clinician diagnosed LN participants.
* At least one visit to the investigational center during 12 months prior to the baseline visit, recorded in medical documentation.
* Literacy in English or Arabic allowing to fully comprehend the written informed consent and study-specific patient reported questionnaires.

Exclusion Criteria:

* Incomplete medical records to be able to assess the disease severity or absence of any of the following renal laboratory results from the medical record within the last twelve months: a. Urinary protein to creatinine ratio (UPCR) or 24-hour proteinuria or urine sediment (activity). b. Serum creatinine or estimated glomerular filtration rate (eGFR); or measured glomerular filtration rate (GFR), if eGFR is not available.
* Current or medical history of: a. Congenital or acquired immunodeficiency. b. Malignancy in active treatment phase. c. Acute viral infection, such as human immunodeficiency virus (HIV) infection, requiring hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with lupus nephritis as defined by physician per participants hospital records prior to the enrolment visit or at diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- GSK Investigational Site, Shweikh, Kuwait
- GSK Investigational Site, Bawshar, Oman
- GSK Investigational Site, Alrayyan, Qatar
- United Arab Emirates (3):
  - GSK Investigational Site, Abu Dhabi
  - GSK Investigational Site, Al Ain City
  - GSK Investigational Site, Dubai

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter prospective study. A total of 193 participants were enrolled in the study.
Groups:
- Participants With Lupus Nephritis: Participants with lupus nephritis as defined by physician per participant hospital records prior to the enrollment visit or at diagnosis were included in this study. No study treatment was administered during conduct of this study.
Period: Overall Study
Arm/Group | Participants With Lupus Nephritis
Started | 193
Completed | 193
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Arab | 164
  Asian | 24
  Black/African-American | 2
  Caucasian/White | 1
  Iranian/Persian | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Categorized by Demographic Characteristics
Description: Number of participants categorized by demographic characteristics including - health insurance coverage (yes, no), employment status (full time, part-time, housewife, not working, other, retired, self-employment), cigarette smoking status (current smoker, ex-smoker, non-smoker, unknown) and alcohol consumption (current, former, never, unknown) has been presented.
Time Frame: At Baseline (Day 1)
Population: "All Subjects Enrolled (ASE) Population" included all participants who met the inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Participants
  Health insurance coverage, yes | 143
  Health insurance coverage, no | 50
  Employment status, full time | 88
  Employment status, part-time | 3
  Employment status, housewife | 30
  Employment status, not working | 58
  Employment status, other | 9
  Employment status, retired | 4
  Employment status, self-employment | 1
  Cigarette smoking status, current smoker | 8
  Cigarette smoking status, ex-smoker | 6
  Cigarette smoking status, non-smoker | 164
  Cigarette smoking status, unknown | 15
  Alcohol consumption, current | 1
  Alcohol consumption, former | 1
  Alcohol consumption, never | 163
  Alcohol consumption, unknown | 28

2. Primary Outcome: Number of Participants With Active Clinical Manifestations of Lupus Nephritis
Description: The active clinical manifestations included pedal edema, serositis, hair loss, decreased urine output, malar rash, discoid rash, photosensitive rash, joint pain/arthritis, hypertension, oral ulcer, seizure, psychosis, proteinuria, microscopic hematuria, anemia, thrombocytopenia, renal failure, leukopenia, other (autoimmune hepatitis, raised Serum creatinine with estimated glomerular filtration rate [eGFR] 59 milliliters per minute [ml/min]/1.73 meter square [m^2]). Participants may have more than 1 active clinical manifestations of Lupus Nephritis.
Time Frame: Up to 12 months
Population: ASE Population. Only those participants who were analyzed (i.e., contributed to data reported in the table) for this outcome measure were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Participants
  Pedal edema | 59
  Serositis | 23
  Hair loss | 46
  Decreased urine output | 13
  Malar rash | 32
  Discoid rash: number analyzed (Participants) | 192
  Discoid rash | 17
  Photosensitive rash: number analyzed (Participants) | 192
  Photosensitive rash | 25
  Joint pain/arthritis | 94
  Hypertension | 64
  Oral ulcer | 21
  Seizure | 9
  Psychosis | 4
  Proteinuria: number analyzed (Participants) | 186
  Proteinuria | 133
  Microscopic hematuria: number analyzed (Participants) | 176
  Microscopic hematuria | 93
  Anemia: number analyzed (Participants) | 192
  Anemia | 81
  Thrombocytopenia: number analyzed (Participants) | 192
  Thrombocytopenia | 24
  Renal failure | 22
  Leukopenia: number analyzed (Participants) | 191
  Leukopenia | 59
  other (autoimmune hepatitis, raised Serum creatinine with eGFR 59 ml/min/1.73m^2) | 2

3. Primary Outcome: Number of Participants With Comorbidities
Description: Participants with comorbidities (such as antiphospholipid syndrome/thrombotic microangiopathy, obesity, cardiovascular disease, diabetes) observed since the date of first diagnosis of lupus nephritis has been presented.
Time Frame: Up to 12 months
Population: "ASE Population" included all participants who met the inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Participants | 134

4. Primary Outcome: Number of Participants With Severe Lupus Nephritis
Description: Severe lupus nephritis was defined as participants with Systemic lupus erythematosus disease activity index 2000 (SLEDAI-2K) score greater than or equal to (>=) 10. SLEDAI-2K score was the sum of all 24 individual items from the SLEDAI-2K. The total score ranges from 0 (no disease activity) to 105 (all 24 descriptors present simultaneously). A higher score indicates a more significant degree of disease activity.
Time Frame: Up to 12 months
Population: ASE Population. Only those participants who were analyzed (i.e., contributed to data reported in the table) for this outcome measure were included in the 'Overall Number of Participants Analyzed' field. Participants with at least one SLEDAI-2K score assessment were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 190
Participants | 60

5. Primary Outcome: Number of Participants Categorized by Treatments for Lupus Nephritis
Description: Number of participants categorized by treatments for lupus nephritis including prednisone, chloroquine, hydroxychloroquine, azathioprine, belimumab, tacrolimus, cyclosporine, voclosporin, cyclophosphamide, mycophenolate mofetil, methotrexate, and rituximab has been presented. Participants may have received more than 1 treatment for lupus nephritis.
Time Frame: At Baseline (Day 1)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Participants
  Prednisone | 152
  Chloroquine: number analyzed (Participants) | 191
  Chloroquine | 2
  Hydroxychloroquine: number analyzed (Participants) | 192
  Hydroxychloroquine | 185
  Azathioprine: number analyzed (Participants) | 192
  Azathioprine | 81
  Belimumab: number analyzed (Participants) | 192
  Belimumab | 19
  Tacrolimus: number analyzed (Participants) | 191
  Tacrolimus | 26
  Cyclosporine: number analyzed (Participants) | 191
  Cyclosporine | 6
  Voclosporin: number analyzed (Participants) | 191
  Voclosporin | 0
  Cyclophosphamide: number analyzed (Participants) | 189
  Cyclophosphamide | 26
  Mycophenolate mofetil: number analyzed (Participants) | 192
  Mycophenolate mofetil | 133
  Methotrexate: number analyzed (Participants) | 189
  Methotrexate | 6
  Rituximab: number analyzed (Participants) | 191
  Rituximab | 27

6. Primary Outcome: Short Form Health Survey (SF-36) Health-related Quality of Life Domain Score
Description: The 36-Item Short Form Health Survey (SF-36) is a 36-item Health-Related Quality of Life (HRQoL) questionnaire covering 8 health domains: physical functioning, Pain, Role limitations due to physical health, Role limitations due to emotional problems, emotional well-being, Social Functioning, energy/fatigue, and General Health. The individual question items are first summed for each item under the various sections. Then, those domain scores were weighted to a scale ranging between 0 to 100, where higher score represents better health. Individual domain scores have been presented.
Time Frame: At Baseline (Day 1)
Population: "ASE Population" included all participants who met the inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Scores on a scale
  Physical functioning | 67.6 (26.9)
  Pain | 59.5 (29)
  Role limitation due to physical health | 64.1 (41.4)
  Role limitation due to emotional problems | 66.5 (41.5)
  Emotional well-being | 67.9 (21.9)
  Social functioning | 69.7 (28.1)
  Energy/fatigue | 57.7 (21.3)
  General health | 49.7 (38.4)

7. Secondary Outcome: Number of Participants With Refractory Lupus Nephritis
Description: Refractory systemic lupus nephritis was defined as inefficacy of cyclophosphamide, use of rituximab, splenectomy, or inefficacy of >=2 immunosuppressives (methotrexate, leflunomide, abatacept, anti-tumor necrosis factor [anti-TNF], azathioprine, mycophenolate mofetil, and/or mycophenolic acid).
Time Frame: Up to 12 months
Population: ASE Population. Only those participants who were analyzed (i.e., contributed to data reported in the table) for this outcome measure were included in the 'Overall Number of Participants Analyzed' field.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 191
Participants | 33

8. Secondary Outcome: Number of Participants With Abnormal Findings for Serological Markers
Description: Number of participants with abnormal findings for serological markers (including anti-nuclear antibody, anti-double-stranded deoxyribonucleic acid [dsDNA] antibody and complement levels [C3, C4]) has been presented. Abnormal values were determined by the investigator.
Time Frame: At 3, 6, 9 and 12 months
Population: "ASE Population" included all participants who met the inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Participants
  Anti-nuclear antibody: at 3 months | 2
  Anti-nuclear antibody: at 6 months | 0
  Anti-nuclear antibody: at 9 months | 2
  Anti-nuclear antibody: at 12 months | 3
  Anti-dsDNA antibody: at 3 months | 52
  Anti-dsDNA antibody: at 6 months | 55
  Anti-dsDNA antibody: at 9 months | 46
  Anti-dsDNA antibody: at 12 months | 56
  C3: at 3 months | 47
  C3: at 6 months | 46
  C3: at 9 months | 42
  C3: at 12 months | 43
  C4: at 3 months | 29
  C4: at 6 months | 28
  C4: at 9 months | 19
  C4: at 12 months | 23

9. Secondary Outcome: Number of Participants With Renal Remission That Were Associated With Clinical Factors, Biomarkers, and Treatments
Description: Renal remission was defined as proteinuria of <0.7 grams per day (g/d) or <0.5g/d or at physicians' discretion. Number of participants with renal remission that were associated with clinical factors, biomarkers, and treatments has been presented.
Time Frame: Up to 12 months
Population: "ASE Population" included all participants who met the inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Participants | 123

10. Secondary Outcome: Percent Change From Baseline in SF-36 Scores for Each Health Domain:Physical Functioning, Pain, Role Limitations Due to Physical Health, Role Limitations Due to Emotional Problem, Emotional Well-being, Social Functioning, Energy/Fatigue and General Health
Description: The 36-Item Short Form Health Survey (SF-36) is a 36-item HRQoL questionnaire covering 8 health domains: physical functioning, pain, role limitations due to physical health, role limitations due to emotional problems, emotional well-being, social functioning, energy/fatigue, and general Health. The individual question items are first summed for each item under the various sections. Then, those domain scores were weighted to a scale ranging between 0 to 100, where higher score represents better health. Baseline was considered as Day 1. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value (at 12 months). Percent change from Baseline was calculated by dividing change from Baseline value by Baseline value and multiplying it by 100. Percent change from Baseline values of individual domain scores have been presented.
Time Frame: Baseline (Day 1) and at 12 months
Population: "ASE Population" included all participants who met the inclusion and exclusion criteria.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Percent change
  Physical functioning | 23.7 (182.5)
  Pain | 29 (126.4)
  Role limitations due to physical health | 1.4 (79.4)
  Role limitations due to emotional problems | 0.9 (69.1)
  Emotional well-being | 6.6 (63.4)
  Social functioning | 13.4 (68.7)
  Energy/fatigue | 11.1 (63.9)
  General health | -2.8 (40.2)

11. Secondary Outcome: Number of Participants With Hospitalizations and Intensive Care Unit (ICU) Hospitalizations
Description: Number of participants with hospitalizations and ICU hospitalizations has been presented.
Time Frame: Up to 12 months
Population: "ASE Population" included all participants who met the inclusion and exclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Participants
  Participants with hospitalizations | 14
  Participants with ICU hospitalizations | 1

12. Secondary Outcome: Direct Medical Costs Associated With Lupus Nephritis Management
Description: The direct medical costs of hospitalization and ICU hospitalization per participant associated with lupus nephritis management in United States dollars (USD) of United Arab Emirates (UAE), Kuwait, Qatar, and Oman were analyzed. Costs are described in local currency of each country and converted in USD dollars using the average exchange rate for each local currency versus USD in 2023. Direct medical costs associated with lupus nephritis management have been reported as USD.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: USD
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 15
USD
  Hospitalizations: UAE: number analyzed (Participants) | 9
  Hospitalizations: UAE | 517 (193.9)
  ICU hospitalizations: UAE: number analyzed (Participants) | 1
  ICU hospitalizations: UAE | 141.6 (NA) — NA indicates data was not available as standard deviation could not be calculated for a single participant.
  Hospitalizations: Kuwait: number analyzed (Participants) | 0
  ICU hospitalizations: Kuwait: number analyzed (Participants) | 0
  Hospitalizations: Qatar: number analyzed (Participants) | 0
  ICU hospitalizations: Qatar: number analyzed (Participants) | 0
  Hospitalizations: Oman: number analyzed (Participants) | 5
  Hospitalizations: Oman | 467.6 (338.7)
  ICU hospitalizations: Oman: number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Treatment for Lupus Nephritis by Sector (Public or Private Sector)
Description: Number of participants with treatments for lupus nephritis (Prednisone, Chloroquine, Hydroxychloroquine, Azathioprine, Belimumab, Tacrolimus, Cyclosporine A, Voclosporin, Cyclophosphamide, Mycophenolate mofetil, Methotrexate, Rituximab) among physicians in the public and private sectors, respectively has been presented. Data has been presented per treatment received either in public sector or private sector up to 12 months. Participants may have received more than 1 treatment.
Time Frame: Up to 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Lupus Nephritis
Number analyzed (Participants) | 193
Participants
  Prednisone prescribed by physicians in public sector: number analyzed (Participants) | 126
  Prednisone prescribed by physicians in public sector | 102
  Prednisone prescribed by physicians in private sector: number analyzed (Participants) | 67
  Prednisone prescribed by physicians in private sector | 48
  Chloroquine prescribed by physicians in public sector: number analyzed (Participants) | 126
  Chloroquine prescribed by physicians in public sector | 2
  Chloroquine prescribed by physicians in private sector: number analyzed (Participants) | 67
  Chloroquine prescribed by physicians in private sector | 0
  Hydroxychloroquine prescribed by physicians in public sector: number analyzed (Participants) | 126
  Hydroxychloroquine prescribed by physicians in public sector | 118
  Hydroxychloroquine prescribed by physicians in private sector: number analyzed (Participants) | 67
  Hydroxychloroquine prescribed by physicians in private sector | 67
  Azathioprine prescribed by physicians in public sector: number analyzed (Participants) | 126
  Azathioprine prescribed by physicians in public sector | 49
  Azathioprine prescribed by physicians in private sector: number analyzed (Participants) | 67
  Azathioprine prescribed by physicians in private sector | 32
  Belimumab prescribed by physicians in public sector: number analyzed (Participants) | 126
  Belimumab prescribed by physicians in public sector | 9
  Belimumab prescribed by physicians in private sector: number analyzed (Participants) | 67
  Belimumab prescribed by physicians in private sector | 11
  Tacrolimus prescribed by physicians in public sector: number analyzed (Participants) | 126
  Tacrolimus prescribed by physicians in public sector | 19
  Tacrolimus prescribed by physicians in private sector: number analyzed (Participants) | 67
  Tacrolimus prescribed by physicians in private sector | 7
  Cyclosporine A prescribed by physicians in public sector: number analyzed (Participants) | 126
  Cyclosporine A prescribed by physicians in public sector | 5
  Cyclosporine A prescribed by physicians in private sector: number analyzed (Participants) | 67
  Cyclosporine A prescribed by physicians in private sector | 1
  Voclosporin prescribed by physicians in public sector: number analyzed (Participants) | 126
  Voclosporin prescribed by physicians in public sector | 0
  Voclosporin prescribed by physicians in private sector: number analyzed (Participants) | 67
  Voclosporin prescribed by physicians in private sector | 0
  Cyclophosphamide prescribed by physicians in public sector: number analyzed (Participants) | 126
  Cyclophosphamide prescribed by physicians in public sector | 19
  Cyclophosphamide prescribed by physicians in private sector: number analyzed (Participants) | 67
  Cyclophosphamide prescribed by physicians in private sector | 7
  Mycophenolate mofetil prescribed by physicians in public sector: number analyzed (Participants) | 126
  Mycophenolate mofetil prescribed by physicians in public sector | 86
  Mycophenolate mofetil prescribed by physicians in private sector: number analyzed (Participants) | 67
  Mycophenolate mofetil prescribed by physicians in private sector | 55
  Methotrexate prescribed by physicians in public sector: number analyzed (Participants) | 126
  Methotrexate prescribed by physicians in public sector | 5
  Methotrexate prescribed by physicians in private sector: number analyzed (Participants) | 67
  Methotrexate prescribed by physicians in private sector | 1
  Rituximab prescribed by physicians in public sector: number analyzed (Participants) | 126
  Rituximab prescribed by physicians in public sector | 20
  Rituximab prescribed by physicians in private sector: number analyzed (Participants) | 67
  Rituximab prescribed by physicians in private sector | 12

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events were collected up to 12 months
Description: All-cause mortality and serious adverse events were collected for ASE Population. Only All-cause mortality and SAEs were collected during the study to comply with regulations of the local authorities. Non-SAEs were not collected in this non interventional study as safety was not a study objective per protocol.
Arm/Group | Participants With Lupus Nephritis
All-Cause Mortality (participants affected / at risk) | 1/193
Serious Adverse Events (participants affected / at risk) | 5/193
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Lupus Nephritis (N=193)
Palpitations (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 1
COVID-19 virus test positive (Infections and infestations) | 1
SLE (Immune system disorders) | 1
Dyspnoea (Immune system disorders) | 1
Influenzal pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Knee pain (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Healthcare Resource Utilization and costs:

1. Relevant data was collected in local currency, as United States Dollar and local currency were used based on a fixed annual rate.
2. In order to map the costs at Government hospitals, these hospitals were asked to list the costs of their services and to describe consultation fees of their salaried healthcare practitioners.
3. Assumptions were made on out-of-pocket expenses that were not recorded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT04971590/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT04971590/SAP_001.pdf